CLINICAL TRIAL: NCT01437137
Title: The Clinical Efficacy of Recently Developed Supraglottic Airway Device, I-gel™, in Neonates and Infants: Comparison With Classic-laryngeal Mask Airway (c-LMA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 1-2011-0052
Record Dates: First submitted 2011-09-14; First posted 2011-09-20 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Airway Complication of Anaesthesia
Keywords: elective surgery of short duration (less than 2 hr) undergoing general anesthesia using supraglottic airway

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- LMA group (Active Comparator)
  Interventions: Device: classic-laryngeal mask airway (c-LMA)
- I-gel group (Experimental)
  Interventions: Device: i-gel™

INTERVENTIONS:
Device: classic-laryngeal mask airway (c-LMA) — Insertion of c-LMA
  Arms: LMA group
Device: i-gel™ — Insertion of I-gel
  Arms: I-gel group

SUMMARY:
Although the safety and efficacy of the Classic-laryngeal mask airway (c-LMA) in children has been shown in several large observational studies, findings suggest that the smaller-sized c-LMAs, in particular sizes 1 and 1½, are less suitable for airway maintenance under general anesthesia in small infants and that they may even be associated with more frequent complications than with the facemask and endotracheal tube. The pediatric i-gel is a new supraglottic airway device for children. It is made of a soft, gel-like elastomer with a noninflatable cuff. Studies about I-gel in adults have been promising, showing an easy insertion, high airway leak pressures, and low complication rates with few postoperative complaints. The aim of this study is to compare clinical performance of the pediatric i-gel and c-LMA in infants.

ELIGIBILITY:
Inclusion Criteria:

* infants (0-1 year of age)
* who scheduled for elective surgery of short duration (less than 2 hr) undergoing general anesthesia using supraglottic airway

Exclusion Criteria:

* patients with an abnormal airway
* with reactive airway disease
* with gastroesophageal reflux disease
* with chronic respiratory disease
* has a history of an upper respiratory tract infection in the preceding 6-week period

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
airway leak pressure | within 5 min of insertion of each device
  Airway leak pressure was determined by adjusting the expiratory valve of the breathing circle to 40 cmH2O (fixed fresh gas flow 3 L/min) and recording the pressure when equilibrium was reached.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Beylacq L, Bordes M, Semjen F, Cros AM. The I-gel, a single-use supraglottic airway device with a non-inflatable cuff and an esophageal vent: an observational study in children. Acta Anaesthesiol Scand. 2009 Mar;53(3):376-9. doi: 10.1111/j.1399-6576.2008.01869.x. PMID 19243322